CLINICAL TRIAL: NCT05114395
Title: Comparison Between a Telerehabilitation Program for Urinary Incontinence Versus a Conventional Face-to-face Program: a Longitudinal Study in Pandemic Times
Brief Title: Comparison Between a Telerehabilitation Program for Urinary Incontinence Versus a Conventional Face-to-face Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar De São João, E.P.E. (Other)
Responsible Party: Principal Investigator, Susana Moreira, Medical Doctor, Centro Hospitalar De São João, E.P.E.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE 114-21
Record Dates: First submitted 2021-05-26; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Stress Urinary Incontinence; Incontinence, Urinary; Covid19; Pelvic Floor Muscle Weakness
Keywords: Pelvic floor; Physical therapy; Urinary incontinence; Quality of life; Telerehabilitation; Training; Pelvic floor musculature; Female; Pelvic Floor Muscle Training
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence; COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Group (Experimental): The intervention group includes a hybrid program of face-to-face sessions and video sessions. In the first consultation, a face-to-face one, patients will be instructed with behavioral and lifestyle measures and it will be prescribed a 12-week exercise program, including exercises to be performed three times a day and two weekly exercise sessions - three face-to-face sessions (2 initial and one at 8 weeks) and video sessions of 30 minutes, divided into 3 phases with gradual addition of exercises of increasing difficulty in terms of duration, number of repetitions and positions.
  In the middle of the treatment (at 6 weeks) a medical teleconsultation is performed for reassessment. In the end of the 12-week program there will also be a face-to-face consultation.
  Interventions: Other: Pelvic Floor Telerehabilitation Program
- Face-to-Face Group (Active Comparator): The control group develops the entire program in face-to-face consultations and exercise sessions.
  Interventions: Other: Pelvic Floor Face-to-Face Program

INTERVENTIONS:
Other: Pelvic Floor Telerehabilitation Program — See experimental and active comparator arms.
  Arms: Telerehabilitation Group
Other: Pelvic Floor Face-to-Face Program — See experimental and active comparator arms.
  Arms: Face-to-Face Group

SUMMARY:
Urinary incontinence (UI) is defined as any involuntary loss of urine. It affects a significant percentage of the population, mainly female, with a prevalence of 21.4% in Portuguese women, having a negative impact on quality of life and sexual function.

About half presents with stress UI (SUI), followed by mixed UI (MUI), with isolated urgency UI being less common.

Pelvic floor rehabilitiation is a first line treatment for SUI and MUI, however, it is not yet defined which is the best treatment program or the ideal strategies to improve adherence to it.

Telerehabilitation assumed a leading role in the covid pandemic phase, although there are few studies on pelvic floor rehabilitation for UI, none in Portugal to date.

The authors aim to evaluate the effectiveness of a hybrid program of pelvic floor rehabilitation in female patients with SUI and MUI with a predominance of SUI, including consultation and face-to-face sessions complemented with telerehabilitation.

DETAILED DESCRIPTION:
Randomized longitudinal study including consecutively admitted patients on pelvic floor rehabilitation consultation of the Physical Medicine and Rehabilitation Department of Centro Hospitalar São João for conservative treatment of UI.

Patients who meet the inclusion criteria and do not meet any of the exclusion criteria will be randomized one to one between the intervention group and the control group.

The intervention group includes a hybrid program of face-to-face sessions followed by sessions of video, while the control group develops the entire program in face-to-face sessions.

The effectiveness of the program will be assessed by the results in the UI-related quality of life (primary outcome); UI severity, patient's overall perception of improvement, sexual function, depression/anxiety symptoms and satisfaction and adherence to treatment (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged between 18 and 65 years with SUI or MUI with a predominance of SUI with at least 1 urinary incontinence episode per week in the last month
* Pelvic floor muscle strength greater than or equal to 2 (modified Oxford scale)
* Capable of understanding and executing the therapeutic program and expressing agreement to participate in the study after free and informed consent

Exclusion Criteria:

* Patients with urgency urinary incontinence or MUI with a predominance of urgency
* Pregnant women
* Submitted to conservative or surgical treatment of UI in the last 12 months
* Active urinary tract infection
* Macroscopic hematuria
* Neurogenic dysfunction of the lower urinary tract
* Cognitive deficit
* Osteoarticular, neurological or psychiatric pathologies that prevent the realization of the therapeutic program
* Active pelvic neoplasia
* Pelvic organ prolapse grade greater than or equal to 2
* Impossibility of access or illiteracy to technological means (phone or computer)
* Unavailable to attend the face-to-face program due to accessibility, schedule, economic reasons or fear of the pandemic context

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 39 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-08-09 (Actual)

PRIMARY OUTCOMES:
Assessment of urinary incontinence related quality of life using the Portuguese Version of the King's Health Questionnaire (KHQ). | From admission to discharge of the program, up to 13 weeks.
  The primary outcome is the assessment of urinary incontinence related quality of life using the Portuguese Version of KHQ.

SECONDARY OUTCOMES:
Assessment of UI severity. | From admission to discharge of the program, up to 13 weeks.
  Assessment of UI severity using the International Continence Society (ICS) pad test.
Evaluation of the global perception of improvement of the patient. | From admission to discharge of the program, up to 13 weeks.
  Evaluation of the global perception of improvement of the patient using the Portuguese version of the Patient Global Impression of Improvement (PGI-I) Scale.
  The minimum value is 0 and the maximum is 10. A higher score means a better outcome.
Evaluation of sexual function. | From admission to discharge of the program, up to 13 weeks.
  Evaluation of sexual function using the Portuguese version of the Female Sexual Functioning Index (FSFI)
Assessment of the presence of symptoms of depression/anxiety. | From admission to discharge of the program, up to 13 weeks.
  Assessment of the presence of symptoms of depression/anxiety using the Portuguese version of the Hospital Anxiety & Depression Scale (HADS) questionnaire.
  The minimum value is 0 and the maximum is 21. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.
Assessment of satisfaction with the treatment. | From admission to discharge of the program, up to 13 weeks.
  Assessment of satisfaction with the treatment using the 9-point Likert scale. The minimum value is 1 and the maximum is 9. A higher score means a better outcome.
Assessment of adherence to the treatment. | From admission to discharge of the program, up to 13 weeks.
  Assessment of adherence to the treatment including compliance to the exercise program (number of performed sessions) and to the behavioral measures.
Assessment of UI severity. | From admission to discharge of the program, up to 16 weeks.
  Assessment of UI severity using the Portuguese version of the International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF).

CONTACTS AND LOCATIONS:
Overall Officials: Susana Moreira, Principal Investigator — Centro Hospitalar Universitário São João
Locations (2):
- Portugal (2):
  - Physical and Rehabilitation Medicine Department - Centro Hospitalar Universitário de São João, Porto
  - Susana Cristina Alves Moreira, Porto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] D'Ancona C, Haylen B, Oelke M, Abranches-Monteiro L, Arnold E, Goldman H, Hamid R, Homma Y, Marcelissen T, Rademakers K, Schizas A, Singla A, Soto I, Tse V, de Wachter S, Herschorn S; Standardisation Steering Committee ICS and the ICS Working Group on Terminology for Male Lower Urinary Tract & Pelvic Floor Symptoms and Dysfunction. The International Continence Society (ICS) report on the terminology for adult male lower urinary tract and pelvic floor symptoms and dysfunction. Neurourol Urodyn. 2019 Feb;38(2):433-477. doi: 10.1002/nau.23897. Epub 2019 Jan 25. PMID 30681183
- [Background] Correia S, Dinis P, Rolo F, Lunet N. Prevalence, treatment and known risk factors of urinary incontinence and overactive bladder in the non-institutionalized Portuguese population. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Dec;20(12):1481-9. doi: 10.1007/s00192-009-0975-x. Epub 2009 Aug 14. PMID 19684999
- [Background] Hay-Smith EJ, Bo Berghmans LC, Hendriks HJ, de Bie RA, van Waalwijk van Doorn ES. Pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2001;(1):CD001407. doi: 10.1002/14651858.CD001407. PMID 11279716
- [Background] Carrion Perez F, Rodriguez Moreno MS, Carnerero Cordoba L, Romero Garrido MC, Quintana Tirado L, Garcia Montes I. [Telerehabilitation to treat stress urinary incontinence. Pilot study]. Med Clin (Barc). 2015 May 21;144(10):445-8. doi: 10.1016/j.medcli.2014.05.036. Epub 2014 Jul 30. Spanish. PMID 25087210
- [Derived] Santiago M, Cardoso-Teixeira P, Pereira S, Firmino-Machado J, Moreira S. A Hybrid-Telerehabilitation Versus a Conventional Program for Urinary Incontinence: a Randomized Trial during COVID-19 Pandemic. Int Urogynecol J. 2023 Mar;34(3):717-727. doi: 10.1007/s00192-022-05108-6. Epub 2022 May 21. PMID 35596802

DOCUMENTS (1):
  • Informed Consent Form (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/95/NCT05114395/ICF_000.pdf